CLINICAL TRIAL: NCT03511521
Title: Use of Neutral Protamine Hagedorn (NPH) Versus Basal Bolus Insulin for Steroid Induced Hyperglycemia
Brief Title: Use of NPH Versus Basal Bolus Insulin for Steroid Induced Hyperglycemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit sufficient number of patients
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mark E Molitch, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00207079
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Hyperglycemia Steroid-induced; Insulin Resistance, Diabetes
Keywords: steroid; prednisone; methylprednisolone; hyperglycemia; insulin; hypoglycemia
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Hyperglycemia; Hypoglycemia | interventions — Insulin, Isophane; Isophane Insulin, Human; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Intervention Model Description: Patients receiving single dose steroids who become hyperglycemic will be randomized to two treatment arms in a parallel design: (1) NPH added to basal/bolus insulin; (2) increase in doses of basal and bolus insulin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NPH Insulin (Experimental): NPH will be given at the time of steroid administration to the patient in addition to standard basal/bolus insulin the patient may be receiving in the following doses:
  Prednisone Dose (mg/day) - NPH dose (U=Units): 10-20 mg/day - 1.2U (units)/mg; 21-40 mg/day - 0.6U/mg; 41-60 mg/day - 0.45U/mg; 61-80 mg/day - 0.3U/mg; >80 mg/day - no additional NPH. Note that the amounts of NPH are added to each other for the various prednisone doses. For example, a dose of 75 mg/day of prednisone would come out to be (1.2U x 20mg = 24U) + (0.6U x 20mg = 12U) + (0.45U x 20mg = 9U) + 0.3U x 15 mg = 4.5U) for a total of 24 + 12 + 9 + 4.5 = 49.5U of NPH for 75 mg of prednisone.
  Interventions: Drug: NPH Insulin; Drug: glargine; Drug: Insulin Aspart
- Basal/Bolus Insulin (Active Comparator): Basal insulin (glargine) and Bolus insulin (insulin aspart) will be increased (doses given in U [units]/kg) according to the Prednisone dose (mg/day) as follows:
  Prednisone Dose (mg/day) - doses of insulin (U/kg): Prednisone 0 mg - Glargine 0.25U/kg, Bkfst Aspart 0.08U/kg, Lunch Aspart 0.08U/kg, Dinner Aspart - 0.08U/kg; Prednisone 10-20 mg - Glargine 0.25U/kg, Bkfst Aspart 0.1U/kg, Lunch Aspart 0.15U/kg, Dinner Aspart - 0.2U/kg; Prednisone 21-40 mg - Glargine 0.25U/kg, Bkfst Aspart 0.1U/kg, Lunch Aspart 0.2U/kg, Dinner Aspart - 0.25U/kg; Prednisone 41-60 mg - Glargine 0.30U/kg, Bkfst Aspart 0.15U/kg, Lunch Aspart 0.25U/kg, Dinner Aspart - 0.30U/kg; Prednisone 61-80 mg - Glargine 0.30U/kg, Bkfst Aspart 0.15U/kg, Lunch Aspart 0.30U/kg, Dinner Aspart - 0.35U/kg; Prednisone >80 mg - Glargine 0.30U/kg, Bkfst Aspart 0.15U/kg, Lunch Aspart 0.35U/kg, Dinner Aspart - 0.40U/kg.
  Interventions: Drug: glargine; Drug: Insulin Aspart

INTERVENTIONS:
Drug: NPH Insulin — Intermediate acting insulin
  Other Names: Humulin N; Novolin N
  Arms: NPH Insulin
Drug: glargine — basal insulin
  Other Names: Lantus; Basaglar
Drug: Insulin Aspart — prandial insulin
  Other Names: Novolog

SUMMARY:
Glucocorticoids are known to cause an increase in insulin resistance, leading to hyperglycemia, in both diabetic and non-diabetic patients. In both the inpatient and outpatient setting, steroids are used for their anti-inflammatory property to treat a variety of conditions. There is a paucity of information regarding the best way to treat steroid-induced hyperglycemia. In this study we will compare (1) the addition of NPH insulin, an intermediate-acting insulin, given at the time of steroid administration to the patient's standard basal/bolus insulin to (2) modification of the standard basal-bolus insulin regimen which will consist primarily increasing the prandial doses at lunch and supper in order to determine which regimen is superior for glycemic control.

DETAILED DESCRIPTION:
Inpatients who will receive single daily doses of prednisone or methylprednisolone for treatment of their underlying condition and who become hyperglycemic will be eligible. Subjects will be randomized in a 1:1 fashion to one of two arms: (1) to their standard basal bolus insulin the addition of NPH insulin given at the time of the steroid adminstration, adjusting the dose based on the dose of steroid; (2) an increase in the basal and prandial bolus insulin doses based on the dose of steroid. Glycemic control and the incidence of hypoglycemia will be assessed over the first 3 days after initiating these insulin regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving once daily dosing of methylprednisolone or prednisone in a dose of 10 mg/day or greater
* Hyperglycemic (Glucose level > 126 mg/dL)
* Diabetic and nondiabetic patients
* Expected duration of hospital stay and time on steroids >= 3 days
* Patient of appropriate caregiver able to give Informed Consent

Exclusion Criteria:

* Patients with 2 or more doses of methylprednisolone/prednisone per day
* Steroids other than methylprednisolone or prednisone
* Pregnancy
* estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Molitch, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dhital SM, Shenker Y, Meredith M, Davis DB. A retrospective study comparing neutral protamine hagedorn insulin with glargine as basal therapy in prednisone-associated diabetes mellitus in hospitalized patients. Endocr Pract. 2012 Sep-Oct;18(5):712-9. doi: 10.4158/EP11371.OR. PMID 22784834
- [Result] Ruiz de Adana MS, Colomo N, Maldonado-Araque C, Fontalba MI, Linares F, Garcia-Torres F, Fernandez R, Bautista C, Olveira G, de la Cruz JL, Rojo-Martinez G, Valdes S. Randomized clinical trial of the efficacy and safety of insulin glargine vs. NPH insulin as basal insulin for the treatment of glucocorticoid induced hyperglycemia using continuous glucose monitoring in hospitalized patients with type 2 diabetes and respiratory disease. Diabetes Res Clin Pract. 2015 Nov;110(2):158-65. doi: 10.1016/j.diabres.2015.09.015. Epub 2015 Sep 30. PMID 26474657
- [Result] Radhakutty A, Stranks JL, Mangelsdorf BL, Drake SM, Roberts GW, Zimmermann AT, Stranks SN, Thompson CH, Burt MG. Treatment of prednisolone-induced hyperglycaemia in hospitalized patients: Insights from a randomized, controlled study. Diabetes Obes Metab. 2017 Apr;19(4):571-578. doi: 10.1111/dom.12859. Epub 2017 Feb 17. PMID 27995731
- [Result] Bevier WC, Zisser HC, Jovanovic L, Finan DA, Palerm CC, Seborg DE, Doyle FJ 3rd. Use of continuous glucose monitoring to estimate insulin requirements in patients with type 1 diabetes mellitus during a short course of prednisone. J Diabetes Sci Technol. 2008 Jul;2(4):578-83. doi: 10.1177/193229680800200408. PMID 19885233
- [Result] Seggelke SA, Gibbs J, Draznin B. Pilot study of using neutral protamine Hagedorn insulin to counteract the effect of methylprednisolone in hospitalized patients with diabetes. J Hosp Med. 2011 Mar;6(3):175-6. doi: 10.1002/jhm.874. No abstract available. PMID 21387555

RESULTS

PARTICIPANT FLOW:
Groups:
- NPH Insulin: NPH will be given at the time of steroid administration to the patient in addition to standard basal/bolus insulin the patient may be receiving in the following doses:
  Prednisone Dose (mg/day) - NPH dose (U=Units): 10-20 mg/day - 1.2U (units)/mg; 21-40 mg/day - 0.6U/mg; 41-60 mg/day - 0.45U/mg; 61-80 mg/day - 0.3U/mg; >80 mg/day - no additional NPH. Note that the amounts of NPH are added to each other for the various prednisone doses. For example, a dose of 75 mg/day of prednisone would come out to be (1.2U x 20mg = 24U) + (0.6U x 20mg = 12U) + (0.45U x 20mg = 9U) + 0.3U x 15 mg = 4.5U) for a total of 24 + 12 + 9 + 4.5 = 49.5U of NPH for 75 mg of prednisone.
  NPH Insulin: Intermediate acting insulin
  glargine: basal insulin
  Insulin Aspart: prandial insulin
- Basal/Bolus Insulin: Basal insulin (glargine) and Bolus insulin (insulin aspart) will be increased (doses given in U [units]/kg) according to the Prednisone dose (mg/day) as follows:
  Prednisone Dose (mg/day) - doses of insulin (U/kg): Prednisone 0 mg - Glargine 0.25U/kg, Bkfst Aspart 0.08U/kg, Lunch Aspart 0.08U/kg, Dinner Aspart - 0.08U/kg; Prednisone 10-20 mg - Glargine 0.25U/kg, Bkfst Aspart 0.1U/kg, Lunch Aspart 0.15U/kg, Dinner Aspart - 0.2U/kg; Prednisone 21-40 mg - Glargine 0.25U/kg, Bkfst Aspart 0.1U/kg, Lunch Aspart 0.2U/kg, Dinner Aspart - 0.25U/kg; Prednisone 41-60 mg - Glargine 0.30U/kg, Bkfst Aspart 0.15U/kg, Lunch Aspart 0.25U/kg, Dinner Aspart - 0.30U/kg; Prednisone 61-80 mg - Glargine 0.30U/kg, Bkfst Aspart 0.15U/kg, Lunch Aspart 0.30U/kg, Dinner Aspart - 0.35U/kg; Prednisone >80 mg - Glargine 0.30U/kg, Bkfst Aspart 0.15U/kg, Lunch Aspart 0.35U/kg, Dinner Aspart - 0.40U/kg.
  glargine: basal insulin
  Insulin Aspart: prandial insulin
Period: Overall Study
Arm/Group | NPH Insulin | Basal/Bolus Insulin
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NPH Insulin | Basal/Bolus Insulin | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (1.5) | 36 (0) | 50.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3
Initial Glucose [Mean (Standard Deviation); unit: mg/dL] | 244 (4) | 80 (0) | 189 (77.4)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control
Description: mean of 4 glucose levels per day (premeal and bedtime) for each group for first 3 days after intervention
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | NPH Insulin | Basal/Bolus Insulin
Number analyzed (Participants) | 2 | 1
mg/dL | 284.3 (81.0) | 184.3 (61.8)

2. Secondary Outcome: Percentage of Glucose Values Within Therapeutic Range
Description: Percentage of the glucose values (premeal and bedtime for 3 days) within the therapeutic target of 80 - 180 mg/dL
Time Frame: 3 days
Measure: Mean (95% Confidence Interval); unit: percentage of glucose values in range
Arm/Group | NPH Insulin | Basal/Bolus Insulin
Number analyzed (Participants) | 2 | 1
percentage of glucose values in range | 4.2 [3.4 to 5.0] | 50 [19 to 81]

3. Secondary Outcome: Percentage of Glucose Values Within the Hypoglycemic Range
Description: Percentage of the glucose values (premeal and bedtime for 3 days) less than 70 mg/dL and 54 mg/dL
Time Frame: 3 days
Measure: Mean (95% Confidence Interval); unit: Percentage of glucose values < 70 mg/dL
Arm/Group | NPH Insulin | Basal/Bolus Insulin
Number analyzed (Participants) | 2 | 1
Percentage of glucose values < 70 mg/dL | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | NPH Insulin | Basal/Bolus Insulin
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03511521/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT03511521/ICF_001.pdf